CLINICAL TRIAL: NCT03550456
Title: Diagnostics of the Quality of Life With Exercise Induced Asthma (EIA) and Exercise Induced Laryngeal Obstruction (EILO)
Brief Title: Diagnostics and Quality of Life With EIA and EILO
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Johannes Schulze MD, Prof., Johann Wolfgang Goethe University Hospital
Other Study IDs: KGU-83/18
Record Dates: First submitted 2018-05-23; First posted 2018-06-08 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Exercise Induced Asthma; Exercise Induced Pharyngeal Collapse
Keywords: Exercise Induced Asthma (EIA); Exercise Induced Laryngeal Obstruction (EILO); Quality of life; Exercise challenge in cold chamber (ECC); Continous laryngoscopy while exercising (CLE)
MeSH Terms: conditions — Asthma, Exercise-Induced | interventions — Eukaryotic Initiation Factor-2B; Speech Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECC, ECC with CLE, speech therapy: After the standard diagnostic (spirometry, body plethysmography, exhaled NO, skin prick test) all patients with dyspnea while exercising undergo exercise challenges in a cold chamber (ECC).
  In case of a positive reaction in the ECC the patients get asthma medication (ICS/LABA combination).
  Both groups negative and positive should fill out a symptom diary and the next visit will be booked 6 weeks later.
  If they still have dyspnea while exercising with ICS/LABA combination or hat a negative ECC the patients undergo an ECC with continuous laryngoscopy. In case of an EILO diagnosis patients will be sent to speech therapy and checked at a follow up visit.
  All patients and their parents should complete questionnaires for symptoms and quality of life at every visit.
  Interventions: Other: ECC; Other: ECC with CLE; Other: Speech therapy

INTERVENTIONS:
Other: ECC — Exercise challenge is defined as running on a treadmill for 6-8 minutes on submaximal work load in a cold chamber.
Other: ECC with CLE — Continuous Laryngoscopy is endoscopy of the larynx used to obtain a view of laryngeal obstruction during exercise.
Other: Speech therapy — Patients with diagnosis of EILO will be sent to a speech therapist for at least 6 training sessions.

SUMMARY:
The purpose of this study is to investigate the quality of life of subjects suffering from dyspnoea while exercising and quantify the number of diagnoses of Exercise induced Asthma (EIA) and Exercise induced laryngeal obstruction (EILO) in our outpatient clinic using an exercise-challenge in a cold-chamber and an exercise-challenge with continuous laryngoscopy.

DETAILED DESCRIPTION:
In this study investigators want to characterize and investigate the quality of life of all patients consulting the outpatient clinic for pediatric pulmonology suffering from dyspnoea while exercising.

Besides standard diagnostics (bodyplethysmograph, spirometry, exhaled NO, skin prick test) subjects will take part in an exercise-challenge in a cold chamber at 2-4°C. Subjects showing symptoms of exercise-induced asthma will get a treatment with ICS/LABA for six weeks. All Patients should fill out a symptom diary. On suspicion of an EILO, subjects not showing symptoms in the first exercise-challenge in the cold chamber and all subjects without improvement after EIA treatment will take part in a second exercise-challenge in the cold chamber with continuous laryngoscopy.

If EILO is proved by laryngoscopy, speech therapy is recommended. To investigate the symptoms and the quality of life of these patients, all patients and there parents should answer symptom and quality of life questionnaires (Child Behavior Checklist (CBCL/4-18), Youth Self-Report (YSR 11-18), Asthma Control Test, (ACT) Dyspnea Index (DI)) at every visit.

There are yearly follow ups of these patients for five years in order to collect long-range prognosis.

ELIGIBILITY:
Inclusion Criteria:

* written agreement
* age: >=8 and <= 18
* exercise induced dyspnea
* at least two training session per week
* lung function before physical exercise FVC >= 75% and FEV1 >= 70%

Exclusion Criteria:

* age <8 and >18
* lung function: forced vital capacity (FVC) < 75% and forced expiratory pressure in one second (FEV1) < 70%
* inability to understand the range oft the study
* chronic asthma with systemic cortisone therapy
* chronic asthma with high dose cortisone inhalation >500 micrograms fluticasone equivalent
* intake of long acting beta-agonists (LABA) 48 h before examination
* acute severe infection (pneumonia) within the last 4 weeks
* intake of leukotriene-antagonists 48h before examination
* other chronic diseases or infections (HIV, Tbc)
* pregnancy

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients from our outpatient clinic aged 8-18 years with exercise induced dyspnea and at least two training session per week.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of life in subjects with exercise induced asthma and exercise induced laryngeal obstruction | 5 years
  The primary endpoint is the quality of life of all subjects with EIA and EILO assessed by questionnaires (Child Behavior Checklist (CBCL/4-18) for parents and Youth Self-Report (YSR 11-18) for adolescents) at the time of diagnosis and after therapy in accordance with the diagnosis with ICS/LABA combination or speech therapy. Both questionnaires are almost identical and contain 120 items (CBCL/4-18) and 119 items (YSR), respectively, in eight different categories: anxious/depressed, withdrawn/depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behavior, and aggressive behavior. Answers to each item are coded on a 3-point Likert-scale, 0 = not true, 1 = somewhat or sometimes true, 2 = very true or often true. Raw scores are transformed into T-scores to allow comparison with children from the same gender and age.

SECONDARY OUTCOMES:
Symptoms of EIA and EILO | 5 years
  Comparison of symptom score ACT and DI between EIA and EILO.
Prevalence | 1 year
  Patients suffering from exercise induced dyspnea are evaluated of prevalence of EIA-, EILO and combinations of EIA+EILO.
Speech therapy | 5 years
  Success monitoring of speech therapy of EILO or combination of EIA+EILO on the basis of a survey concerning the quality of life and symptoms.
Carbon dioxide | 5 years
  Changes in the concentration of carbon dioxide in the blood by capillary blood gas analysis before and after the exercise challenge in a cold chamber and before and after CLE diagnostics.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Schulze, Assoc. Prof., Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (1):
- Goethe University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Parsons JP, Hallstrand TS, Mastronarde JG, Kaminsky DA, Rundell KW, Hull JH, Storms WW, Weiler JM, Cheek FM, Wilson KC, Anderson SD; American Thoracic Society Subcommittee on Exercise-induced Bronchoconstriction. An official American Thoracic Society clinical practice guideline: exercise-induced bronchoconstriction. Am J Respir Crit Care Med. 2013 May 1;187(9):1016-27. doi: 10.1164/rccm.201303-0437ST. PMID 23634861
- [Background] Anderson SD, Charlton B, Weiler JM, Nichols S, Spector SL, Pearlman DS; A305 Study Group. Comparison of mannitol and methacholine to predict exercise-induced bronchoconstriction and a clinical diagnosis of asthma. Respir Res. 2009 Jan 23;10(1):4. doi: 10.1186/1465-9921-10-4. PMID 19161635
- [Background] Driessen JM, van der Palen J, van Aalderen WM, de Jongh FH, Thio BJ. Inspiratory airflow limitation after exercise challenge in cold air in asthmatic children. Respir Med. 2012 Oct;106(10):1362-8. doi: 10.1016/j.rmed.2012.06.017. Epub 2012 Jul 11. PMID 22789953
- [Background] Maat RC, Roksund OD, Halvorsen T, Skadberg BT, Olofsson J, Ellingsen TA, Aarstad HJ, Heimdal JH. Audiovisual assessment of exercise-induced laryngeal obstruction: reliability and validity of observations. Eur Arch Otorhinolaryngol. 2009 Dec;266(12):1929-36. doi: 10.1007/s00405-009-1030-8. Epub 2009 Jul 8. PMID 19585139
- [Background] Schulze J, Smith HJ, Fuchs J, Herrmann E, Dressler M, Rose MA, Zielen S. Methacholine challenge in young children as evaluated by spirometry and impulse oscillometry. Respir Med. 2012 May;106(5):627-34. doi: 10.1016/j.rmed.2012.01.007. Epub 2012 Feb 10. PMID 22326606
- [Background] Schulze J, Rosewich M, Riemer C, Dressler M, Rose MA, Zielen S. Methacholine challenge--comparison of an ATS protocol to a new rapid single concentration technique. Respir Med. 2009 Dec;103(12):1898-903. doi: 10.1016/j.rmed.2009.06.007. Epub 2009 Jul 10. PMID 19596563
- [Background] Schulze J, Rosewich M, Dressler M, Riemer C, Rose MA, Zielen S. Bronchial allergen challenge using the Medicaid dosimeter. Int Arch Allergy Immunol. 2012;157(1):89-97. doi: 10.1159/000324473. Epub 2011 Sep 7. PMID 21912178
- [Background] Schulze J, Voss S, Zissler U, Rose MA, Zielen S, Schubert R. Airway responses and inflammation in subjects with asthma after four days of repeated high-single-dose allergen challenge. Respir Res. 2012 Sep 19;13(1):78. doi: 10.1186/1465-9921-13-78. PMID 22989372
- [Background] Roksund OD, Heimdal JH, Clemm H, Vollsaeter M, Halvorsen T. Exercise inducible laryngeal obstruction: diagnostics and management. Paediatr Respir Rev. 2017 Jan;21:86-94. doi: 10.1016/j.prrv.2016.07.003. Epub 2016 Jul 18. PMID 27492717
- [Background] Buchvald F, Phillipsen LD, Hjuler T, Nielsen KG. Exercise-induced inspiratory symptoms in school children. Pediatr Pulmonol. 2016 Nov;51(11):1200-1205. doi: 10.1002/ppul.23530. Epub 2016 Sep 22. PMID 27717246
- [Background] Johansson H, Norlander K, Berglund L, Janson C, Malinovschi A, Nordvall L, Nordang L, Emtner M. Prevalence of exercise-induced bronchoconstriction and exercise-induced laryngeal obstruction in a general adolescent population. Thorax. 2015 Jan;70(1):57-63. doi: 10.1136/thoraxjnl-2014-205738. Epub 2014 Nov 7. PMID 25380758
- [Background] Nielsen EW, Hull JH, Backer V. High prevalence of exercise-induced laryngeal obstruction in athletes. Med Sci Sports Exerc. 2013 Nov;45(11):2030-5. doi: 10.1249/MSS.0b013e318298b19a. PMID 23657163
- [Background] Heimdal JH, Roksund OD, Halvorsen T, Skadberg BT, Olofsson J. Continuous laryngoscopy exercise test: a method for visualizing laryngeal dysfunction during exercise. Laryngoscope. 2006 Jan;116(1):52-7. doi: 10.1097/01.mlg.0000184528.16229.ba. PMID 16481809
- [Background] Christensen PM, Thomsen SF, Rasmussen N, Backer V. Exercise-induced laryngeal obstructions: prevalence and symptoms in the general public. Eur Arch Otorhinolaryngol. 2011 Sep;268(9):1313-9. doi: 10.1007/s00405-011-1612-0. Epub 2011 Apr 29. PMID 21528411
- [Background] Christensen PM, Maltbaek N, Jorgensen IM, Nielsen KG. Can flow-volume loops be used to diagnose exercise induced laryngeal obstructions? A comparison study examining the accuracy and inter-rater agreement of flow volume loops as a diagnostic tool. Prim Care Respir J. 2013 Sep;22(3):306-11. doi: 10.4104/pcrj.2013.00067. PMID 23955336